CLINICAL TRIAL: NCT06903234
Title: Post-authorization Safety Study of Iptacopan in Adult Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH) Using Data From the Non-interventional IPIG PNH Registry
Brief Title: Post-authorization Safety Study of Iptacopan in Adult Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH) Using Data From the IPIG PNH Registry
Status: Active, not recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLNP023C12003
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Hemoglobinuria, Paroxysmal
Keywords: Paroxysmal nocturnal hemoglobinuria; Iptacopan
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — iptacopan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Iptacopan: Adult patients with PNH treated with iptacopan in routine care.
  Interventions: Drug: Iptacopan

INTERVENTIONS:
Drug: Iptacopan — Adult patients with PNH treated with iptacopan
  Other Names: Fabhalta

SUMMARY:
This is an observational single-arm descriptive cohort study based on the secondary use of data collected on iptacopan-treated patients with paroxysmal nocturnal hemoglobinuria (PNH) through the International PNH Interest Group (IPIG) PNH registry.

DETAILED DESCRIPTION:
This multinational, non-interventional, descriptive single-arm cohort study is based on secondary analysis of data collected within the iptacopan silo of the IPIG PNH Registry (data on iptacopan-treated patients made available to Novartis). This is a non-interventional study utilizing secondary data and is considered a "registry-based study." The IPIG PNH Registry (CT.gov NCT06524726), the parent registry, includes a dedicated drug silo to collect data from patients using iptacopan in routine care.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent to participate in the IPIG PNH Registry
* PNH confirmed by flow cytometry
* Incident users of iptacopan
* Aged at least 18 years at the iptacopan initiation

Exclusion Criteria:

* Participation in an interventional clinical trial

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with PNH who are enrolled in the IPIG PNH Registry, newly treated with iptacopan.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2029-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with infections caused by encapsulated bacteria | From initiation of iptacopan until discontinuation + 3 days, or end of follow-up, up to 5 years.
  To describe the risk of infections caused by encapsulated bacteria in patients with PNH treated with iptacopan in routine clinical practice. Infections caused by encapsulated bacteria (Neisseria meningitidis, Streptococcus pneumoniae, Haemophilus influenzae).
Cumulative incidence of infections (event probability as a function of time), caused by encapsulated bacteria | From initiation of iptacopan until discontinuation + 3 days, or end of follow-up, up to 5 years.
  To describe the risk of infections caused by encapsulated bacteria in patients with PNH treated with iptacopan in routine clinical practice. Infections caused by encapsulated bacteria (Neisseria meningitidis, Streptococcus pneumoniae, Haemophilus influenzae).
Number of patients with infections events per 100 participants -years (incidence rates) caused by encapsulated bacteria | From initiation of iptacopan until discontinuation + 3 days, or end of follow-up, up to 5 years.
  To describe the risk of infections caused by encapsulated bacteria in patients with PNH treated with iptacopan in routine clinical practice. Infections caused by encapsulated bacteria (Neisseria meningitidis, Streptococcus pneumoniae, Haemophilus influenzae).
Number of infections episodes per 100 patients -years (occurrence rates) caused by encapsulated bacteria | From initiation of iptacopan until discontinuation + 3 days, or end of follow-up, up to 5 years.
  To describe the risk of infections caused by encapsulated bacteria in patients with PNH treated with iptacopan in routine clinical practice. Infections caused by encapsulated bacteria (Neisseria meningitidis, Streptococcus pneumoniae, Haemophilus influenzae).

SECONDARY OUTCOMES:
Number of patients with serious infections caused by encapsulated bacteria and all serious infection | From initiation of iptacopan until discontinuation + 3 days, or end of follow-up, up to 5 years.
  To describe the short- and long-term risk of the serious infections in patients with PNH treated with iptacopan in routine clinical practice. Infections caused by encapsulated bacteria (Neisseria meningitidis, Streptococcus pneumoniae, Haemophilus influenzae) and all serious infection.
Cumulative incidence of serious infections, caused by encapsulated bacteria and all serious infection (event probability as a function of time) | From initiation of iptacopan until discontinuation + 3 days, or end of follow-up, up to 5 years.
  To describe the short- and long-term risk of the serious infections in patients with PNH treated with iptacopan in routine clinical practice. Infections caused by encapsulated bacteria (Neisseria meningitidis, Streptococcus pneumoniae, Haemophilus influenzae) and all serious infection.
Number of patients with serious infections events per 100 patients -years (incidence rates) caused by encapsulated bacteria and all serious infection | From initiation of iptacopan until discontinuation + 3 days, or end of follow-up, up to 5 years.
  To describe the short- and long-term risk of the serious infections in patients with PNH treated with iptacopan in routine clinical practice. Infections caused by encapsulated bacteria (Neisseria meningitidis, Streptococcus pneumoniae, Haemophilus influenzae) and all serious infection.
Number of serious infections episodes per 100 patients -years (occurrence rates) caused by encapsulated bacteria and all serious infection | From initiation of iptacopan until discontinuation + 3 days, or end of follow-up, up to 5 years.
  To describe the short- and long-term risk of the serious infections in patients with PNH treated with iptacopan in routine clinical practice. Infections caused by encapsulated bacteria (Neisseria meningitidis, Streptococcus pneumoniae, Haemophilus influenzae) and all serious infection.
Number of patients with potential breakthrough hemolysis, solid tumors, hematological malignancies, Major adverse vascular events (MAVEs), serious adverse events (SAEs), hyperlipidemia and thrombocytopenia | From initiation of iptacopan until discontinuation + 3 days, or end of follow-up, up to 5 years.
  To describe the short- and long-term risk of potential breakthrough hemolysis, solid tumors, hematological malignancies, MAVEs, SAEs, hyperlipidemia and thrombocytopenia in patients with PNH treated with iptacopan in routine clinical practice.
Cumulative incidence of potential breakthrough hemolysis, solid tumors, hematological malignancies, MAVEs, SAEs, hyperlipidemia and thrombocytopenia (event probability as a function of time) | From initiation of iptacopan until discontinuation + 3 days, or end of follow-up, up to 5 years.
  To describe the short- and long-term risk of potential breakthrough hemolysis, solid tumors, hematological malignancies, MAVEs, SAEs, hyperlipidemia and thrombocytopenia in patients with PNH treated with iptacopan in routine clinical practice.
Number of patients with potential breakthrough hemolysis, solid tumors, hematological malignancies, MAVEs, SAEs, hyperlipidemia and thrombocytopenia events per 100 patients -years (incidence rates) | From initiation of iptacopan until discontinuation + 3 days, or end of follow-up, up to 5 years.
  To describe the short- and long-term risk of potential breakthrough hemolysis, solid tumors, hematological malignancies, MAVEs, SAEs, hyperlipidemia and thrombocytopenia in patients with PNH treated with iptacopan in routine clinical practice.
Number of potential breakthrough hemolysis, solid tumors, hematological malignancies, MAVEs, SAEs, hyperlipidemia and thrombocytopenia episodes per 100 patients -years (occurrence rates) | From initiation of iptacopan until discontinuation + 3 days, or end of follow-up, up to 5 years.
  To describe the short- and long-term risk of potential breakthrough hemolysis, solid tumors, hematological malignancies, MAVEs, SAEs, hyperlipidemia and thrombocytopenia in patients with PNH treated with iptacopan in routine clinical practice.
Number of patients with death due to any cause | From initiation of iptacopan until discontinuation + 3 days, or end of follow-up, up to 5 years.
  To describe the short- and long-term risk of all-cause mortality in patients with PNH treated with iptacopan in routine clinical practice.
Cumulative incidence of death due to any cause (event probability as a function of time) | From initiation of iptacopan until discontinuation + 3 days, or end of follow-up, up to 5 years.
  To describe the short- and long-term risk of all-cause mortality in patients with PNH treated with iptacopan in routine clinical practice.
Number of patients with death due to any cause events per 100 patients -years (incidence rates) | From initiation of iptacopan until discontinuation + 3 days, or end of follow-up, up to 5 years.
  To describe the short- and long-term risk of all-cause mortality in patients with PNH treated with iptacopan in routine clinical practice.
Number of patients vaccinated against Neisseria meningitidis, Streptococcus pneumoniae, Haemophilus influenzae at each study visit | From initiation of iptacopan until discontinuation + 3 days, or end of follow-up, up to 5 years.
  To describe the number of patients receiving mandatory and recommended vaccinations against encapsulated bacteria.
Number of patients with serious hemolysis following discontinuation of iptacopan | From the iptacopan discontinuation up to 14 days
  To describe the risk of serious hemolysis following discontinuation of iptacopan in patients with PNH treated with iptacopan in routine clinical practice.
Number of patients who became pregnant during treatment with iptacopan, exposure characteristics (e.g. trimester of exposure) and birth outcomes | From the Last Menstrual Period to pregnancy outcome (in case of live birth, up to 12 months post delivery)
  To describe the frequency of use of iptacopan during pregnancy in PNH patients, characteristics of pregnancies exposed to iptacopan and frequency of selected pregnancy and birth outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Novartis Investigative Site, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No